CLINICAL TRIAL: NCT01556529
Title: CDRM Study: Computer-assisted Diabetes Risk Management-evaluation of a Medical Care Approach to Support Secondary and Tertiary Prevention of Type 2 Diabetes Mellitus and Its Complications
Brief Title: CDRM Study: Computer-assisted Diabetes Risk Management-for Secondary and Tertiary Prevention of T2DM Complications
Acronym: CDRM_DMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Prof. Ulrich Mueller, PROFESSOR, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDRM 92/07/56
Record Dates: First submitted 2012-02-21; First posted 2012-03-16 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- risk profile information (Experimental): patient gets information on quantitative individual complication risk profile and patient gets standard T2DM DMP care
  Interventions: Procedure: risk profile information; Procedure: standard DMP care
- Control (Active Comparator): Control group: patient gets standard T2DM DMP care
  Interventions: Procedure: standard DMP care

INTERVENTIONS:
Procedure: risk profile information — (1) patient on a regular basis receives individualized reports on his/her quantitative risk for 6 typical diabetes complications over the next 10 years, (2) standard T2DMP care, as outlined by AWMF diabetes guidelines
  Other Names: risk calculator
  Arms: risk profile information
Procedure: standard DMP care — standard disease management of T2DM care
  Other Names: AWMF Guidelines oriented care
  Arms: Control
Procedure: standard DMP care — standard disease management of T2DM care
  Other Names: risk calculator
  Arms: risk profile information

SUMMARY:
The CDRM study will evaluate a newly developed approach to improve management and secondary prevention in diabetes care. The research will explore the impact of an medical care intervention via a computer-assisted diabetes risk management system (CDRMS) on compliance and outcome The focus will be on the effect on patients' diabetes and diabetes complication risk profiles, medical effectiveness and patients- reported outcomes.

DETAILED DESCRIPTION:
The study will determine the effects of a computer-assisted diabetes risk management (CDRM) system on compliance and outcome. All subjects are Type 2 Diabetes Mellitus (T2DM) patients enrolled in the National T2DM Disease Management Programme (DMP) offered by the German National Health Insurance System. Of all people living in Germany 90% are insured there; more than 60% of all T2DM patients insured there are - voluntarily - enrolled in the T2DM-DMP. As in any DMP, the rationale is that by regular visits to the attending physician, strict application of National Guidelines and by keeping the patient in a narrow corridor of optimal biomedical parameters (SBP, DBP, BMI, and specific lab parameters), the probability of complications, hospitalizations and other functional impairments is minimized.

The rationale of the study is that more information on individual risk profile and its changes in the course of care will lead to more patient empowerment adding to more effective preventing the manifestation of these risks.

The Intervention Group, in addition to receiving the T2DM care standard according to the National Guidelines issued by AWMF, within the framework of the National T2DM Disease Management Programme, will receive individualized reports showing their personal risk for the characteristic T2DM complications. Reports are sent to attending general practitioners (GP) for communicating and explaining them to patients.

The CDRM system entails a combination of several telematic instruments used by the patient, GP and medical specialists. Key functionalities of the network supporting the care approach are the software integration of GP practices and an automated data recording via digital devices of blood glucose meters. Furthermore, the CDRM-Tool, Accu-Chek Mellibase a client server application of Roche Diagnostics GmbH is connected to the system.

It generates reports - one for the physician and one for the patient - on the current health status, describing the 10 year risk to develop a characteristic complication (separately for myocardial infarction, stroke, kidney failure, blindness, amputation) and the potential to reduce this risk. These reports shall be used during consultations to help doctors and patients to communicate about diabetes associated risks and individual potential. The GP report shall ease doctor's therapy decisions. The patient report shall inform the patient to improve compliance, strengthen empowerment. The CDRM system gains this information by correlating the basic patient data plus the data from recent medical findings with the most recent diabetes research evidence. GPs of this intervention group will only get advice concerning how to use the CDRM system properly, no further (extra) intervention measures are permitted. In particular, no therapy recommendations from the research team to GPs how to decide on individual therapy or medication.

The control group will receive the T2DM care standard according to the National Guidelines issued by AWMF, within the framework of the National T2DM Disease Management Programme.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM,
* Enrollment in a T2DM RSAV DMP (German State Health Insurance DMP)

Exclusion Criteria:

* Pregnant
* Dementia, psychoses, or other illness that would hinder compliance
* Serious illness such as:

  * cancer,
  * immune deficiency syndrome (HIV),
  * genetic lipid disorder (e.g. autosomal dominant familial hypercholesteremia).
* Malabsorption syndromes such as colitis and Morbus Crohns disease.
* Bed-ridden or required supportive care
* Cardiac insufficiency > NYHA class II
* Chronic metabolic storage illnesses such as Morbus Wilson or Amyloidosis.
* Endocrinologic diseases with elevated anti-insulin hormone (e.g. hyperthyreosis, pheochromocytoma, acromegaly.
* Chronic inflammatory diseases.
* Chronic therapy with corticosteroids, diazoxide.
* Pancreatic Diabetes mellitus (e.g. alcoholism, chronic pancreatitis, pancreatic resection)
* Any illness that would prevent the active involvement of the patient in the present study
* Prevalence of diabetes typical complications

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
HbA1c, incidence of typical diabetes complications | 36 months (max)

SECONDARY OUTCOMES:
quantitative diabetes typical complication risk profile | 36 months (max)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich O Mueller, MD PhD, Principal Investigator — Medical School, Marburg University, Marburg, State of Hesse: Germany
Locations (1):
- Philipps University Marburg Medical Center, Marburg, Germany

REFERENCES:
- See also: Deutsches Register Klinischer Studien (German Clinical Trials Register) — http://www.drks.de